CLINICAL TRIAL: NCT05929066
Title: A Master Protocol to Investigate the Efficacy and Safety of LY3437943 Once Weekly in Participants Without Type 2 Diabetes Who Have Obesity or Overweight: A Randomized, Double-Blind, Placebo-Controlled Trial (TRIUMPH-1)
Brief Title: A Study of Retatrutide (LY3437943) in Participants Who Have Obesity or Overweight
Acronym: TRIUMPH-1
Status: Active, not recruiting | Phase: Phase 3 | Type: Interventional
Sponsor: Eli Lilly and Company (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 18557; J1I-MC-GZBJ (Other: Master Protocol Eli Lilly and Company); J1I-MC-GOA1 (Other: ISA Eli Lilly and Company); J1I-MC-GSA1 (Other: ISA Eli Lilly and Company); 2023-503657-35-00 (Other: EU Trial Number)
Record Dates: First submitted 2023-06-26; First posted 2023-07-03 (Actual); Last update posted 2025-04-18 (Actual); Status verified 2025-04

CONDITIONS: Obesity; Overweight; Osteoarthritis, Knee; Obstructive Sleep Apnea
MeSH Terms: conditions — Obesity; Overweight; Osteoarthritis, Knee; Sleep Apnea, Obstructive | interventions — retatrutide

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (5):
- Retatrutide Dose 1 (Experimental): Participants will receive retatrutide subcutaneously (SC).
  Interventions: Drug: Retatrutide
- Retatrutide Dose 2 (Experimental): Participants will receive retatrutide SC.
  Interventions: Drug: Retatrutide
- Retatrutide Dose 3 (Experimental): Participants will receive retatrutide SC.
  Interventions: Drug: Retatrutide
- Placebo (Placebo Comparator): Participants will receive placebo.
  Interventions: Drug: Placebo
- Retatrutide Extension Period (Experimental): Participants will receive retatrutide after the placebo-controlled 80 week treatment period for an additional 24 weeks.
  Interventions: Drug: Retatrutide

INTERVENTIONS:
Drug: Retatrutide — Administered SC
  Other Names: LY3437943
  Arms: Retatrutide Dose 1; Retatrutide Dose 2; Retatrutide Dose 3; Retatrutide Extension Period
Drug: Placebo — Administered SC
  Arms: Placebo

SUMMARY:
The purpose of this study is to evaluate the efficacy and safety of retatrutide in participants who have obesity or overweight (J1I-MC-GZBJ master protocol) including subsets of participants who have knee osteoarthritis (OA) (J1I-MC-GOA1) or who have obstructive sleep apnea (OSA) (J1I-MC-GSA1). This study will last about 89 weeks and will include up to 24 visits. Addendum (2) is optional and available to approximately 500 participants to continue treatment with retatrutide for up to an additional 24 weeks.

ELIGIBILITY:
Inclusion Criteria:

* Have body mass index (BMI) ≥30.0 kilograms per square meter (kg/m²), or ≥27.0 kg/m² with at least one of the following:

  * hypertension
  * dyslipidemia
  * obstructive sleep apnea, or
  * cardiovascular disease
* History of of at least one unsuccessful dietary effort to reduce body weight

GOA1 Inclusion Criteria:

* Have index knee pain for >12 weeks prior to screening, and presence of index knee pain for >15 days over the previous month
* Have knee X-ray with moderate radiographic changes (Kellgren-Lawrence Grade 2 or 3) per central reading at screening
* Currently meets American College of Rheumatology (ACR) Criteria (clinical and radiological) for OA.

GSA1 Inclusion Criteria:

* Previously diagnosed with OSA
* Have AHI ≥15 on polysomnography at screening (definition of moderate-to-severe OSA)
* For participants not on positive airway pressure (PAP) therapy: unable or unwilling to use PAP therapy and have not used PAP for at least 4 weeks prior to screening.
* If on PAP therapy, have been on PAP therapy for at least 3 consecutive months prior to screening, and willing to temporarily stop using PAP therapy for approximately 7 days prior to each of the sleep study (PSG) visits.

GZBJ Addenda (2) inclusion criteria:

* Have completed the final treatment visit of GZBJ Week 80.

Exclusion Criteria:

* Have a self-reported or documented change in body weight >5 kg (11 pounds) within 90 days.
* Have taken weight loss drugs, including over-the-counter medications, within 90 days prior to screening.
* Have a prior or planned surgical treatment for obesity.
* Have diabetes mellitus.
* Have family or personal history of medullary thyroid carcinoma (MTC) or multiple endocrine neoplasia syndrome type 2 (MEN-2)
* Have had pancreatitis.

GOA1 exclusion criteria

* Have had steroid joint injections within 90 days of screening.
* Have had other joint injections and procedures within 6 months of screening.
* Have joint disease other than osteoarthritis.

GSA1 exclusion criteria

* Use stimulants (for example, modafinil, armodafinil, solriamfetol, pitolisant, amphetamine) less than 3 months prior to screening.
* Use hypnotics, mirtazapine, opioids, trazodone, and zonisamide less than 3 months prior to screening.
* Use a dental appliance or other device to treat OSA other than PAP therapy.

GZBJ Addenda (2) exclusion criteria

* Have had study intervention discontinuation.
* Have had permanent dose reduction.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 2300 (Estimated)
Dates: Start 2023-07-10 (Actual); Primary Completion 2026-04 (Estimated); Study Completion 2026-05 (Estimated)

PRIMARY OUTCOMES:
Percent Change From Baseline in Body Weight | Baseline, Week 80
Change from Baseline in the Western Ontario and McMaster Universities Osteoarthritis Index (WOMAC) Pain Subscale Score for GOA1 Subset | Baseline, Week 80
Change from Baseline in Apnea-Hypopnea Index (AHI) Events Per Hour for GSA1 Subset | Baseline, Week 80
Percent Change from Baseline in Body Weight to | Baseline, Week 104

SECONDARY OUTCOMES:
Change from Baseline in Body Mass Index (BMI) | Baseline, Week 80
Change from Baseline in Waist Circumference | Baseline, Week 80
Change from Baseline in Systolic Blood Pressure (SBP) | Baseline, Week 80
Percent Change form Baseline in Fasting Insulin | Baseline, Week 80
Change from Baseline in HbA1c | Baseline, Week 80
Change from Baseline in Short Form 36 Version 2 (SF-36v2) Acute Form Physical Functioning Domain Score | Baseline, Week 80
Pharmacokinetics (PK): Steady State Area Under the Concentration Time Curve (AUC) | Baseline through Week 80
  AUC is presented as a single average measure of AUC across the study duration.
Change from Baseline in the WOMAC Physical Function Subscale Score for GOA1 Subset | Baseline, Week 80
Change from Baseline in Average Pain Intensity Numeric Rating Scale (API-NRS) Score for GOA1 Subset | Baseline, Week 80
Change from Baseline in Worst Pain Intensity Numeric Rating Scale (WPI-NRS) Score for GOA1 Subset | Baseline, Week 80
Percent Change from Baseline in AHI for GSA1 Subset | Baseline, Week 80
A Hierarchical Combination of Functional Outcomes of Sleep Questionnaire (FOSQ) 10 Score, FOSQ Vigilance Domain Score, and FOSQ Activity Level Domain Score for GSA1 Subset | Baseline to Week 80
  A hierarchical combination of change from baseline in the FOSQ 10 score, FOSQ Vigilance Domain Score, and FOSQ Activity Level Domain Score will be assessed by the win ratio. The reported unit will be the total "wins" for each treatment group from performing a hierarchical comparison of the components.
Percentage of Participants with ≥50% AHI Reduction from Baseline for GSA1 Subset | Baseline to Week 80
Percentage of Participants with AHI <5 or with AHI 5-14 with Epworth Sleepiness Scale (ESS) ≤10 for GSA1 Subset | Week 80

CONTACTS AND LOCATIONS:
Overall Officials: Call 1-877-CTLILLY (1-877-285-4559 or 1-317-615-4559 Mon - Fri 9 AM - 5 PM Eastern Time (UTC/GMT - 5 hours, EST), Study Director — Eli Lilly and Company
Locations (134):
- United States (39):
  - Central Phoenix Medical Clinic, Phoenix, Arizona
  - Arizona Research Center, Phoenix, Arizona
  - Medical Investigations, Little Rock, Arkansas
  - Neuro-Pain Medical Center, Fresno, California
  - Valley Research, Fresno, California
  - Artemis Institute for Clinical Research, San Diego, California
  - University of Colorado Anschutz Medical Campus, Aurora, Colorado
  - Yale University School of Medicine, New Haven, Connecticut
  - Chase Medical Research, LLC, Waterbury, Connecticut
  - Teradan Clinical Trials, LLC, Brandon, Florida
  - Suncoast Research Group, Miami, Florida
  - New Horizon Research Center, Miami, Florida
  - Clinical Neuroscience Solutions, Orlando, Florida
  - Progressive Medical Research, Port Orange, Florida
  - NeuroTrials Research Inc, Atlanta, Georgia
  - North Georgia Clinical Research, Woodstock, Georgia
  - East-West Medical Research Institute, Honolulu, Hawaii
  - Northwestern University, Chicago, Illinois
  - Central Illinois Diabetes and Clinical Research a Division of Prairie Education and Research Cooperative, Springfield, Illinois
  - Brengle Family Medicine, Indianapolis, Indiana
  - Cotton O'Neil Diabetes & Endocrinology, Topeka, Kansas
  - MedVadis Research Corporation, Waltham, Massachusetts
  - Great Lakes Research Group, Inc., Bay City, Michigan
  - StudyMetrix Research, City of Saint Peters, Missouri
  - Clinvest Research LLC, Springfield, Missouri
  - Palm Research Center Tenaya, Las Vegas, Nevada
  - Rochester Clinical Research, LLC, Rochester, New York
  - Carteret Medical Group, Morehead City, North Carolina
  - Trial Management Associates - Wilmington - Floral Parkway, Wilmington, North Carolina
  - Lillestol Research, Fargo, North Dakota
  - Altoona Center For Clinical Research, Duncansville, Pennsylvania
  - Tribe Clinical Research, LLC, Greenville, South Carolina
  - Tribe Clinical Research - Spartanburg, Spartanburg, South Carolina
  - Vanderbilt Health One Hundred Oaks, Nashville, Tennessee
  - FutureSearch Trials of Neurology, Austin, Texas
  - Juno Research, Houston, Texas
  - Advanced Research Institute, Ogden, Utah
  - Northwest Clinical Research Center, Bellevue, Washington
  - Rainier Clinical Research Center, Renton, Washington
- Australia (8):
  - Emeritus Research, Botany, New South Wales
  - The AIM Centre / Hunter Diabetes Centre, Merewether, New South Wales
  - Logan Hospital, Meadowbrook, Queensland
  - Fusion Clinical Research, Adelaide, South Australia
  - Nightingale Research, Adelaide, South Aust
  - Emeritus Research, Camberwell, Victoria
  - Barwon Health, Geelong, Victoria
  - One Clinical Research, Nedlands, Western Australia
- Brazil (3):
  - CPCLIN, São Paulo, São Paulo
  - CPQuali Pesquisa Clínica, São Paulo
  - CEPIC - Centro Paulista de Investigação Clínica, São Paulo
- Canada (9):
  - Aggarwal and Associates Limited, Brampton, Ontario
  - Dr. Steven V. Zizzo Medicine Professional Corporation, Hamilton, Ontario
  - Wharton Medical Clinic, Hamilton, Ontario
  - Your Research Network, Niagara Falls, Ontario
  - Bluewater Clinical Research Group Inc., Sarnia, Ontario
  - Canadian Phase Onward, Toronto, Ontario
  - Centre de Recherche Clinique de Laval, Laval, Quebec
  - Clinique de médecine Urbaine du Quartier Latin, Montreal, Quebec
  - C.I.C. Mauricie inc., Trois-Rivières, Quebec
- Hungary (8):
  - Szegedi Tudományegyetem Szent-Györgyi Albert Klinikai Központ, Szeged, Csongrád megye
  - Regia Med Kft, Székesfehérvár, Fejér
  - Medifarma 98 Kft, Nyíregyháza, Nyíregyháza
  - DRC Gyógyszervizsgáló Központ, Balatonfüred, Veszprém megye
  - Óbudai Egészségügyi Centrum, Budapest
  - ClinDiab Kft., Budapest
  - Debreceni Egyetem Klinikai Központ, Debrecen
  - Debreceni Egyetem Klinikai Kozpont, Debrecen
- India (14):
  - Endolife Speciality Hospitals, Guntur, Andhra Pradesh
  - Avron Hospitals, Ahmedabad, Gujarat
  - Surat Institute of Digestive Sciences Hospitals, Surat, Gujarat
  - Karnataka Institute of Medical Sciences, Hubli, Karnataka
  - Indian Institute of Diabetes, Thiruvananthapuram, Kerala
  - Jothydev's Diabetes and Research Center, Trivandrum, Kerala
  - Wockhardt Hospital - Mumbai Central, Mumbai, Maharashtra
  - Deenanath Mangeshkar Hospital & Research Centre, Pune, Maharashtra
  - Chellaram Diabetes Institute, Pune, Maharashtra
  - Lifepoint Multispeciality Hospital, Pune, Maharashtra
  - All India Institute of Medical Sciences, Bhubaneswar, Odisha
  - Eternal Heart Care Center and Research Institute, Jaipur, Rajasthan
  - Christian Medical College Vellore, Vellore, Tamil Nadu
  - ILS Hospitals, Kolkata, West Benga
- Mexico (15):
  - Centro de Investigacion en Artritis y Osteoporosis SC, Mexicali, Estado de Baja California
  - Diseno y Planeacion en Investigacion Medica, Guadalajara, Jalisco
  - Clinica de Investigacion en Reumatologia y Obesidad S. C., Guadalajara, Jalisco
  - Private Practice - Dr. Arechavaleta Granell Maria del Rosario, Guadalajara, Jalisco
  - Unidad de Investigación Clínica y Atención Médica HEPA, Guadalajara, Jalisco
  - RM Pharma Specialists, Mexico City, Mexico City
  - Clinica Omega, Mexico City, Mexico City
  - Instituto de Diabetes, Obesidad y Nutricion, Cuernavaca, Morelos
  - Unidad biomedica avanzada monterrey, Monterrey, Nuevo León
  - Hospital Universitario Dr. Jose Eleuterio Gonzalez, Monterrey, Nuevo León
  - EME RED Hospitalaria, Mérida, Yucatán
  - Kohler and Milstein Research S.A. de C.V., Mérida, Yucatán
  - Centro de Atención e Investigación Clínica, Aguascalientes
  - Investigacion En Salud Y Metabolismo S.C / Nutricion Clinica / Unidad de Base de Datos, Chihuahua City
  - Arké SMO S.A de C.V, Veracruz
- Poland (12):
  - Centrum Zdrowia Metabolicznego Pawel Bogdanski, Poznan, Greater Poland Voivodeship
  - INTERCOR, Bydgoszcz, Kuyavian-Pomeranian Voivodeship
  - Private Practice - Dr. Robert Witek, Tarnów, Lesser Poland Voivodeship
  - CenterMed Lublin NZOZ, Lublin, Lublin Voivodeship
  - Gabinety TERPA, Lublin, Lublin Voivodeship
  - MICS Centrum Medyczne Warszawa, Warsaw, Masovian Voivodeship
  - Uniwersytecki Szpital Kliniczny w Białymstoku, Bialystok, Podlaskie Voivodeship
  - Centrum Badan Klinicznych PI-House sp. z o.o., Gdansk, Pomeranian Voivodeship
  - NZOZ Salvia CM, Katowice, Silesian Voivodeship
  - Ambulatorium Sp. z o.o., Elblag, Warmian-Masurian Voivodeship
  - Centrum Kliniczno-Badawcze, Elblag, Warmian-Masurian Voivodeship
  - Specjalistyczna Praktyka Lekarska Diabetologia, Leczenie Cukrzycy i Otylosci, Kielce, Świętokrzyskie Voivodeship
- Ponce Medical School Foundation Inc., Ponce, Puerto Rico
- Romania (10):
  - Diabdana, Oradea, Bihor County
  - C.M.D.T.A. Neomed, Brasov, Brașov County
  - Hightech Medical Services SRL-Centrul pentru Studiul Metabolismului, Bucharest, București
  - Gama Diamed, Mangalia, Constanța County
  - Cabinet Medical Dr.Geru, Timișoara, Timiș County
  - SC Minimed SRL, Bacau
  - Diamed Obesity, Galați
  - Centrul Medical Consultmed, Iași
  - Clinica Korall, Satu Mare
  - Policlinica Astra Sibiu, Sibiu
- Spain (6):
  - CHUAC-Complejo Hospitalario Universitario A Coruña, A Coruña, A Coruña [La Coruña]
  - Complejo Hospitalario Universitario de Ferrol (CHUF)- Hospital Naval, Ferrol, A Coruña [La Coruña]
  - Hospital Universitari Vall d'Hebron, Barcelona, Barcelona [Barcelona]
  - Hospital Universitario Marqués de Valdecilla, Santander, Cantabria
  - Hospital General Universitario de Valencia, Valencia, Valenciana, Comunitat
  - Clínica nuevas Tecnologías en Diabetes y Endocrinología (NTDE), Seville
- United Kingdom (9):
  - Rowden Surgery, Chippenham, England
  - Layton Medical Centre, Blackpool, Lancashire
  - Leicester General Hospital, Leicester, Leicestershire
  - Panthera Biopartners - North London, Enfield, London, City of
  - Glasgow Royal Infirmary, Glasgow, Scotland
  - Heartlands Hospital, Birmingham
  - Aintree University Hospital NHS Foundation Trust, Liverpool
  - St Clare Medical Centre, Penzance
  - Panthera Biopartners - Sheffield, Sheffield

IPD SHARING:
Plan to Share IPD: Yes
Anonymized individual patient level data will be provided in a secure access environment upon approval of a research proposal and a signed data sharing agreement.
Supporting Information: Study Protocol, SAP, CSR
Time Frame: Data are available 6 months after the primary publication and approval of the indication studied in the US and European Union (EU), whichever is later. Data will be indefinitely available for requesting
Access Criteria: A research proposal must be approved by an independent review panel and researchers must sign a data sharing agreement.
URL: http://vivli.org/

REFERENCES:
- See also: A Study of Retatrutide (LY3437943) in Participants Who Have Obesity or Overweight (TRIUMPH-1) — https://trials.lilly.com/en-US/trial/408235